CLINICAL TRIAL: NCT06724289
Title: Psilocybin-Assisted Therapy for Prolonged Grief
Brief Title: Psilocybin for Prolonged Grief Disorder
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jennifer Kim Penberthy, PhD, ABPP, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSR231647
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Prolonged Grief Disorder
Keywords: prolonged grief disorder; psilocybin; psychedlic-assisted treatment; psilocybin-assisted therapy; grief; grief disorder
MeSH Terms: conditions — Prolonged Grief Disorder | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: All eligible participants will receive 25 mg of psilocybin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open-label, single arm trial (Experimental): 25 mg psilocybin administered to each participant
  Interventions: Drug: Psilocybin 25 mg

INTERVENTIONS:
Drug: Psilocybin 25 mg — 25 mg psilocybin administered to each participant in single arm, open-label trial

SUMMARY:
The primary purpose of this study is to explore the feasibility of conducting a clinical trial on the effects of psilocybin for individuals with prolonged grief disorder (PGD).

DETAILED DESCRIPTION:
The study aims to investigate whether a single dose of 25 mg psilocybin can reduce the symptoms of grief and trauma associated with PGD. It is hypothesized that psilocybin will significantly reduce the symptoms of PGD and that the treatment will facilitate subjective mystical, spiritual, or insightful experiences, which in turn may contribute to the alleviation of grief and trauma symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21 years old up to and including 65 years of age
* People of childbearing potential that are sexually active must agree to continue or initiate practice of a highly effective means of birth control, alone or in combination with another, throughout the study. Highly effective options are: implants, intrauterine devices (IUD), and sterilization. Exclusive use of condoms is not effective.
* Negative screen for illicit drugs at first visit
* Consent to all study procedures
* Have an existing diagnosis of Prolonged Grief Disorder
* Agree to abstain from any psychoactive drugs on the day prior to and the day of the drug administration session
* Have low risk for suicidality
* Stable on antidepressant medication for at least two months before screening visit
* Be medically stable as determined by screening for medical problems via a personal interview, a medical questionnaire, a physical examination, an electrocardiogram (ECG), and routine medical blood and urinalysis laboratory tests (CBC, CMP, urine beta-HCG, urine toxicology screen)
* Participant must agree to taper or not consume caffeine on the day of intervention
* Agree not to take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours of each drug administration
* Agree that for one week before each drug session, participant will refrain from taking any nonprescription medication, nutritional supplement, or herbal supplement except when approved by the study investigators. Exceptions will be evaluated by the study investigators and will include acetaminophen, non-steroidal anti-inflammatory drugs (example, Ibuprofen), and common doses of vitamins and minerals
* Have limited lifetime use of hallucinogens
* Willingness and ability to remain within the observation room for the duration of the study drug session, which is up to 10 hours (bathroom breaks are allowed)
* Willingness and ability to follow study protocol as directed by research staff
* Willing and able to attend all sessions in the study and complete follow up assessments
* Fluent in English

Exclusion Criteria:

-General medical exclusion criteria:

* Use of a psychedelic drug within the past 5 years
* Clinically significant transaminitis (AST or ALT greater than two times normal value)
* Person who is pregnant, nursing, or planning to get pregnant determined at screening and before drug session by urine test or self-report
* People of childbearing potential that are sexually active who are not practicing an effective means of birth control
* Cardiovascular conditions: coronary artery disease, stroke, angina, uncontrolled hypertension (identified as >170 systolic or >110 diastolic, on three consecutive readings by study team or study physician's interpretation of health and medication history), a clinically significant ECG abnormality (e.g., atrial fibrillation), prolonged QTc interval (i.e., QTc > 450 msec), heart valve, or TIA in the past year.
* History of head trauma with neurological deficit; seizures, or neurologic disorders including cerebrovascular disease, epilepsy, or neurogenerative diseases
* Type 1 diabetes
* BMI <18
* Currently taking on a regular (e.g., daily) basis any antidepressant medications other than SSRIs, SNRIs, or bupropion, or any other medications that have a primary centrally-acting serotonergic effect, including MAOIs. Bupropion dosage must be < 300 mg in order to be included
* Nicotine dependence that would be incompatible with remaining in study area for the entirety of the 8-10-hour study drug session
* Prescribed or illicit use of benzodiazepines or opioids within 4 weeks prior to screening
* Baseline blood pressure greater than 139/79 (after repeat measures) unless stable with medication as determined by PI or PI designate
* Taking any muscle relaxers, antihistamines, or other medications known to cause lethargy or impair cognitive ability within one day prior to psilocybin session
* Serious medical comorbidity requiring medical intervention or close supervision
* History of claustrophobia
* Any court mandated or legal restrictions that would impair the participant from attending all visits
* Inability to follow and comply with all study procedures
* Deemed unable to meaningfully or safely participate in the study
* Any legal judgement toward subject determined to interfere with study attendance or jeopardize compliance with study protocol determined by PI or designate

General psychiatric exclusion criteria:

* Severe psychiatric disorder (other than depression) within 6 months or lifetime history of serious psychiatric or neurological disorders, including bipolar disorder, or active psychosis
* Clinically significant suicidal ideation (e.g., with strong intent or means) within past 6 months or lifetime history of suicide attempt. ***At any point during the study, a participant may be withdrawn from the study for concerns of suicidality and provided follow-up care by our team or a referral to care if needed.
* Current or past history of meeting criteria for schizophrenia spectrum or other psychotic disorders, or bipolar I disorder
* Current or previous history within one year of meeting criteria for a moderate or severe alcohol, or other drug use disorder (excluding tobacco, caffeine, and cannabis)
* Nicotine dependence that would be incompatible with an individual to be nicotine free for 8-10 hours on a study drug session day
* Have a first degree relative with schizophrenia or other psychotic disorders (except substance/medication-induced or due to another medical condition), or bipolar I disorder

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Aim 1 | From administration of study drug to 6-month follow-up
  To evaluate the feasibility of a single arm, open-label trial design, in which a preparation session will be followed by a single dose of psilocybin 25mg PO in a separate session, followed by two separate semi-structured integration sessions administered to adult participants who meet criteria for prolonged grief disorder. We will conduct 6 months of follow up, measuring recruitment rates and dropout rates, and evaluate the changes in the primary outcome measure of PGD to inform the design of a phase 2 trial.

SECONDARY OUTCOMES:
Aim 2 | Baseline to 6 months after administration of study drug
  2.1. To assess changes over time related to the intervention of the 25 mg of psilocybin and two integration sessions. We hypothesize that the intervention will significantly reduce symptoms of PGD, measured by the Inventory of Complicated Grief (ICG). We will also assess related symptoms of PTSD that typically occur using the Davidson Trauma Scale (DTS) and hypothesize significant reductions in these scores over time as well. Post-treatment assessments will occur immediately after the final session and at 1, 3, and 6-month follow-ups.
  2.2. To evaluate the hypothesis that 25 mg of psilocybin facilitates subjective mystical, spiritual, or insightful experiences that are associated with decreases in grief and trauma symptoms. Participants' experiences will be assessed using the Mystical Experiences Questionnaire, 11-Dimensions of Altered States of Consciousness Questionnaire, the Awe Experience Scale, the Challenging Experiences Questionnaire and the Psychological Insight Questionairre

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Penberthy, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States